CLINICAL TRIAL: NCT03246113
Title: Investigation of Cannabis For Tolerability and Feasibility in Patients Receiving Concurrent Chemoradiation for Glioblastoma.
Brief Title: Tolerability of Cannabis in Patients Receiving Concurrent Chemoradiation for Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of subject interest due to study design
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Margaret Haney, Professor of Neurobiology (in Psychiatry), New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#7290
Record Dates: First submitted 2017-07-25; First posted 2017-08-11 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Glioblastoma
Keywords: GBM WHO Grade IV
MeSH Terms: conditions — Glioblastoma | interventions — nabiximols; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cannabis + Chemoradiation (Experimental): Patients will receive a cannabis strain with high cannabidiol (4.8%) and low Delta-9-THC (3.23%). Patients will smoke the cannabis over a 2 hour session (from 0.5 - 2.0 cannabis cigarettes) before receiving chemoradiation therapy with radiation and concurrent temozolomide.
  Interventions: Drug: Cannabis; Drug: Temozolomide; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Cannabis — Cannabis cigarettes provided by NIDA that contain high levels of CBD (4.8%) and low levels of THC (3.23%). Patients will smoke one-half (1/2) to two (2) cannabis cigarettes prior to receiving chemoradiation.
  Other Names: Marijuana
Drug: Temozolomide — Oral alkylating agent with demonstrated antitumor activity.
Radiation: Radiation Therapy — standard fractionation radiotherapy of 60 Gy in 30 treatments with temozolomide.

SUMMARY:
The goal of this single arm Phase I feasibility study is to investigate the tolerability of cannabis with concurrent chemoradiation in the treatment of glioblastoma multiforme (GBM). A strain of cannabis provided by The National Institute of Drug Abuse (NIDA) that has a high concentration of cannabidiol (CBD) and a low concentration of THC (relative to average street cannabis) will be tested in order to maximize clinical efficacy while minimizing intoxicating side effects in this medically-ill population.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility and the effects of cannabis with high concentrations of CBD in patients receiving chemoradiation for GBM. This is not a therapeutic study for the treatment of glioblastoma. Patients will first complete a cannabis sampling session to assess for initial marijuana tolerability. Proceeding this, patients will complete 3-5 outpatient smoking sessions per week over a 6 week period. During each session, patients will be given 90 minutes to smoke 0.5 to 2 cannabis cigarettes. Outcome measures will include measures of pain, mood, nausea, quality of life, and the both the potentially positive and negative subjective effects of cannabis. Food intake, opioid use, and compliance to cannabis treatment will be investigated. It is hypothesized that concurrent use of cannabis with chemoradiation in the treatment of patients with GBM will be feasible, well tolerated and may decrease radiation-induced toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Glioblastoma requiring standard care chemoradiation of concurrent Temozolomide and 60 Gy of radiation given over 30 treatments
* Age 21-70
* Able to give informed consent, and comply with study procedures

Exclusion Criteria:

* Meet DSM-V criteria for current major psychiatric illness, such as bipolar disorder, major depression, active suicidal intent, or psychosis that could be exacerbated by the administration of cannabis
* Meet DSM-V criteria for major neurological disorder, such as mild cognitive impairment or neurodegenerative disorders (such as movement disorders, dementia), that could be exacerbated by the administration of cannabis.
* Women who are not practicing an effective form of birth control (condoms, diaphragm, birth control pill, IUD) or currently pregnant.
* Current (weekly) use of cannabis.
* Patients on supplemental oxygen or history of chronic obstructive pulmonary disease (COPD).
* Cardiovascular Disease
* Compromised Immunity
* Patients with a history of substance use disorder other than nicotine, such an opiate use disorder.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 6 weeks
  Number of cannabis-related adverse events
  A 44-item computerized subjective-effects questionnaire visual analog scale (VAS), comprising a series of 100-mm lines labeled 'not at all' (0 mm) at one end and 'extremely' at the other end, will be completed at baseline, after the 90 minutes of cannabis availability and at the end of the session. The VAS included mood, physical symptom, and drug effect descriptors; participants will be instructed to rate the extent to which each descriptor applied to them at that moment.

SECONDARY OUTCOMES:
Number of Radiation Induced Toxicities | 6 weeks
  All patients receiving radiation treatments are routinely seen by the radiation oncologist once a week for a status check. The RTOG cooperative group common toxicity criteria will be used to assess for neurological toxicities including paresthesia, weakness, somnolence or agitation, incoordination, headache, hearing deficit, tremor, speech deficit, and ataxia.
Number of Opioid Medications Administered | 6 weeks
  Patients will be asked to provide to us the number of opioid medications they took over the 6-week treatment course. The amount of opioids used will be converted to oral morphine equivalents and tallied for each day.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, PhD, Principal Investigator — Professor of Neurobiology (in Psychiatry) at Columbia University; Tony J Wang, MD, Principal Investigator — Associate Professor of Radiation Oncology at Columbia University Medical Center
Locations (2):
- United States (2):
  - Columbia University Medical Center- Department of Radiation Oncology, New York, New York
  - New York State Psychiatric Institute, New York, New York

IPD SHARING:
Plan to Share IPD: No